CLINICAL TRIAL: NCT04238975
Title: Randomized, Double-blind, Active-controlled Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of GC3111 in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Efficacy(Immunogenicity) of GC3111 in Healthy Adults
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC3111_P2
Record Dates: First submitted 2020-01-08; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Tetanus; Diphtheria; Whooping Cough
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GC3111 Vaccine Group (Experimental): Participants randomized to receive a single dose of GC3111 vaccine (Biological: GC3111 vaccine).
  Interventions: Biological: GC3111 vaccine
- Boostrix® Vaccine Group (Active Comparator): Participants randomized to receive a single dose of Boostrix® vaccine (Biological: Boostrix® vaccine).
  Interventions: Biological: Boostrix® vaccine

INTERVENTIONS:
Biological: GC3111 vaccine — 0.5mL, Intramuscular
  Other Names: GC3111
  Arms: GC3111 Vaccine Group
Biological: Boostrix® vaccine — 0.5mL, Intramuscular
  Other Names: Boostrix®
  Arms: Boostrix® Vaccine Group

SUMMARY:
The purpose of this study is to evaluate safety and efficacy (immunogenicity) of a single dose of GC3111 versus Boostrix® vaccine among healthy adults in 19-64 years of age.

DETAILED DESCRIPTION:
To evaluate immunogenicity of GC3111 as tetanus, diphtheria and acellular pertussis (Tdap) vaccine in healthy adults.

To evaluate safety of GC3111 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged above 19 and under 64 at the time of screening
2. Subject without history of administrating vaccines including diphtheria, tetanus or whooping cough antigens within 2 years prior to administration of investigational drug
3. Subject who provided informed consent and assent forms

Exclusion Criteria:

1. Subject who received vaccine within 4 weeks prior to receiving study vaccine
2. Subject who received Tdap vaccine prior to receiving study vaccine
3. Subject with chronic cough history within 12 weeks before receiving study vaccine
4. Subject who is pregnant, lactating, or of child bearing potential without using an effective method of contraception or not practicing abstinence
5. Subject who participated in any other clinical study (investigational drug/equipment) within 6 months before receiving study vaccine
6. Subject with any condition that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Solicited Adverse Events Following Vaccination with Either GC3111 or Boostrix® Vaccine | Day 0 (pre-vaccination) to Day 14 (post-vaccination)
Unsolicited Adverse Events Following Vaccination with Either GC3111 or Boostrix® Vaccine | Day 0 (pre-vaccination) to Day 28 (post-vaccination)
Serious Adverse Events Following Vaccination with Either GC3111 or Boostrix® Vaccine | Day 0 (pre-vaccination) to Day 180 (post-vaccination)
Vital Signs | Day 0 (pre-vaccination), Day 28 (post-vaccination)
  Blood Pressure (systolic, diastolic) in mmHg
Vital Signs | Day 0 (pre-vaccination), Day 28 (post-vaccination)
  Pulse Rate in pulses per minute
Vital Signs | Day 0 (pre-vaccination), Day 28 (post-vaccination)
  Body Temperature in degrees Celcius
Laboratory Examinations | Screening (pre-vaccination), Day 28 (post-vaccination)
  Blood Test (WBC with differential count (lymphocyte, monocyte etc.), RBC, hemoglobin, hematocrit, platelet count
Laboratory Examinations | Screening (pre-vaccination), Day 28 (post-vaccination)
  Blood Chemistry Test (K, Na, Cl, P, ALT, AST etc.)
Laboratory Examinations | Screening (pre-vaccination), Day 28 (post-vaccination)
  Urine Test (pH, specific gravity, bilirubin etc.)

SECONDARY OUTCOMES:
Ratio of Participants with Antibody Responses (Seroprotection rate) to Tetanus and Diphtheria Components Following Vaccination With Either GC3111 or Boostrix® Vaccine | Day 0 (pre-vaccination) to Day 28 (post-vaccination)
Ratio of Participants With Antibody Responses (Boosting Response rate) to Tetanus and Diphtheria Components Following Vaccination With Either GC3111 or Boostrix® Vaccine | Day 0 (pre-vaccination) to Day 28 (post-vaccination)
Geometric Mean Concentrations (GMC) for Diphtheria, Tetanus and Acellular Pertussis Antigens | Day 28 (post-vaccination)
Geometric Mean Ratio (GMR) of Post-vaccination versus Pre-vaccination antibody concentrations for Diphtheria, Tetanus and Acellular Pertussis Antigens | Day 0 (pre-vaccination) to Day 28 (post-vaccination)

OTHER OUTCOMES:
Functional Antibody Response of Pertussis | Day 0 (pre-vaccination) to Day 28 (post-vaccination)
Stratified Analysis of Pertussis according to Anti-Pertussis antibody titer (Positive/Negative) | Day 0 (pre-vaccination), Day 28 (post-vaccination)

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic Univ. of Korea Eunpyeong St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No